CLINICAL TRIAL: NCT02981459
Title: Pilot Study: Mirabegron for the Treatment of Pain Motivated Urinary Frequency and Urgency in Women, an Open Label Study With Dose Escalation
Brief Title: Mirabegron for the Treatment of Pain Motivated Urinary Frequency and Urgency in Women
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawn by Sponsor
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Tova Ablove, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030-586061
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Urinary Frequency/Urgency; Bladder Irritable; Bladder Pain Syndrome
Keywords: bladder pain; urinary frequency; urinary urgency; mirabegron
MeSH Terms: conditions — Urinary Bladder, Overactive; Cystitis, Interstitial | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mirabegron 25 mg or 50 mg (Experimental)
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — daily mirabegron 25mg with the option to increase dose based on symptoms to 50mg daily after 4 weeks
  Other Names: Myrbetriq

SUMMARY:
The specific purpose of this study is to provide objective data in prospective open label design (n=40) to support the use of Mirabegron as a treatment for pain related urinary frequency and urgency. Women with bladder pain have a poor response to traditional anticholinergic therapy for their symptoms of frequency and urgency.

DETAILED DESCRIPTION:
Hypothesis: Mirabegron is effective in reducing symptoms in women with pain related urinary frequency and urgency.

Specific Aims:

1. To measure the efficacy of Mirabegron in the treatment of frequency and urgency, using voiding diaries.
2. To measure the number of patients with a 50% or greater reduction in frequency and urgency, using voiding diaries.
3. To measure the number of patients with a 50% or greater reduction in bladder pain as measured in the O'Leary-Sant (OLS) IC symptom and problem, and the Lowell Parsons Pelvic Pain and Urgency/Frequency (PUF) patient symptom scale.

Intervention/Project goal: Treatment with Mirabegron 25mg for 4 weeks with an option for dose escalation to 50mg. Duration of study 12 weeks.

Inclusion criteria: Women between the ages of 18 and 89 with complaints of pain related urinary frequency are eligible to participate in the study.

Exclusion criteria:

Patients will be excluded from the study if they have:

1. Severe Liver disease, Child-Pugh class c
2. Severe Kidney disease, GFR<30
3. Elevated blood pressure > 160/95 (in package insert bp >180/110)
4. Urinary retention
5. Pregnant, will become pregnant, or are nursing
6. History of recurrent urinary tract infection
7. Tachycardia: pulse > 100
8. Presently on study drug mirabegron; patient must be willing to participate in a 30 day washout period to be eligible for inclusion
9. Medications - metoprolol, desipramine, digoxin, propafenone, thioridazine, flecainide, warfarin

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking women
2. Age: 18 and 89 years
3. Pain related urinary frequency or urgency associated with >70% of voids. With a minimum of 7 pain motivated voids in 24 hours.
4. Bladder capacity: > 300 ml
5. Urinary frequency: 10 or more voids in 24/hours on voiding diary

Exclusion Criteria:

1. Severe Liver disease: Child-Pugh class c
2. Severe Kidney disease: GFR<30
3. Elevated blood pressure > 160/95 (in package insert bp >180/110)
4. Pregnant, will become pregnant, or are nursing during the study
5. History of recurrent urinary tract infection: 3 or more culture proven urinary tract infections in the past 12 months. An active urinary tract infection.
6. Tachycardia: pulse > 100, or any other history of arrhythmia
7. Intense urge: bladder volumes of <150 ml on cystometry
8. Presently on study drug mirabegron; patient must be willing to participate in a 30 day washout period to be eligible for inclusion
9. Medications: metoprolol, desipramine, digoxin, propafenone, thioridazine, flecainide, warfarin
10. Pain medications: no dose changes in narcotic or non-steroidal medications while on study. Patient must be on a stable medication dose for at least 30 days prior to the screening visit.
11. Neurogenic pain medications such as gabapentin or amitriptyline: no dose changes while on study. Patient must be on a stable medication dose for at least 30 days prior to the screening visit.
12. Anticholinergic medications for incontinence: no dose changes while on study. Patient must be on a stable medication dose for at least 30 days prior to the screening visit.

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The number of pain motivated voids per 24 hours. | 12 weeks

SECONDARY OUTCOMES:
The mean change from baseline to end of study in the daily average number of voids | 12 weeks
The Mean change in global urinary symptoms based upon scores from the Urgency Severity and Impact Questionnaire (USIQ) | 12 weeks
The mean change in the Patient Perception of Bladder Condition (PPBC) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tova S Ablove, MD, Principal Investigator — University at Buffalo; Vanessa Barnabei, MD PHD, Study Chair — University at Buffalo
Locations (1):
- UBMD Obstetrics and Gynecology, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, van Kerrebroeck P, Victor A, Wein A. The standardisation of terminology of lower urinary tract function: report from the Standardisation Sub-committee of the International Continence Society. Am J Obstet Gynecol. 2002 Jul;187(1):116-26. doi: 10.1067/mob.2002.125704. No abstract available. PMID 12114899
- [Background] Aizawa N, Homma Y, Igawa Y. Effects of mirabegron, a novel beta3-adrenoceptor agonist, on primary bladder afferent activity and bladder microcontractions in rats compared with the effects of oxybutynin. Eur Urol. 2012 Dec;62(6):1165-73. doi: 10.1016/j.eururo.2012.08.056. Epub 2012 Sep 5. PMID 22981677
- [Background] Aizawa N, Igawa Y, Nishizawa O, Wyndaele JJ. Effects of CL316,243, a beta 3-adrenoceptor agonist, and intravesical prostaglandin E2 on the primary bladder afferent activity of the rat. Neurourol Urodyn. 2010 Jun;29(5):771-6. doi: 10.1002/nau.20826. PMID 19816919
- [Background] Geoffrion R; UROGYNAECOLOGY COMMITTEE. Treatments for overactive bladder: focus on pharmacotherapy. J Obstet Gynaecol Can. 2012 Nov;34(11):1092-1101. doi: 10.1016/S1701-2163(16)35440-8. PMID 23231848
- [Background] Hood B, Andersson KE. Common theme for drugs effective in overactive bladder treatment: inhibition of afferent signaling from the bladder. Int J Urol. 2013 Jan;20(1):21-7. doi: 10.1111/j.1442-2042.2012.03196.x. Epub 2012 Oct 17. PMID 23072271
- [Background] Irwin DE, Milsom I, Hunskaar S, Reilly K, Kopp Z, Herschorn S, Coyne K, Kelleher C, Hampel C, Artibani W, Abrams P. Population-based survey of urinary incontinence, overactive bladder, and other lower urinary tract symptoms in five countries: results of the EPIC study. Eur Urol. 2006 Dec;50(6):1306-14; discussion 1314-5. doi: 10.1016/j.eururo.2006.09.019. Epub 2006 Oct 2. PMID 17049716
- [Background] Michel MC. beta-Adrenergic Receptor Subtypes in the Urinary Tract. Handb Exp Pharmacol. 2011;(202):307-18. doi: 10.1007/978-3-642-16499-6_15. PMID 21290233
- [Background] Miki T, Matsunami M, Nakamura S, Okada H, Matsuya H, Kawabata A. ONO-8130, a selective prostanoid EP1 receptor antagonist, relieves bladder pain in mice with cyclophosphamide-induced cystitis. Pain. 2011 Jun;152(6):1373-1381. doi: 10.1016/j.pain.2011.02.019. Epub 2011 Mar 10. PMID 21396778
- [Background] Milsom I, Abrams P, Cardozo L, Roberts RG, Thuroff J, Wein AJ. How widespread are the symptoms of an overactive bladder and how are they managed? A population-based prevalence study. BJU Int. 2001 Jun;87(9):760-6. doi: 10.1046/j.1464-410x.2001.02228.x. PMID 11412210
- [Background] Stewart WF, Van Rooyen JB, Cundiff GW, Abrams P, Herzog AR, Corey R, Hunt TL, Wein AJ. Prevalence and burden of overactive bladder in the United States. World J Urol. 2003 May;20(6):327-36. doi: 10.1007/s00345-002-0301-4. Epub 2002 Nov 15. PMID 12811491
- [Background] Yoshimura N, Seki S, Chancellor MB, de Groat WC, Ueda T. Targeting afferent hyperexcitability for therapy of the painful bladder syndrome. Urology. 2002 May;59(5 Suppl 1):61-7. doi: 10.1016/s0090-4295(01)01639-9. PMID 12007524